CLINICAL TRIAL: NCT06674616
Title: Achieving Cardiovascular Health Equity in Community Mental Health: Optimizing Implementation Strategies: An Implementation Trial
Brief Title: Achieving Cardiovascular Health Equity in Community Mental Health: Optimizing Implementation Strategies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00410086; UH3HL154280 (NIH)
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Risk Factors; Serious Mental Illness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Replicating Effective Programs (REP) (Active Comparator)
  Interventions: Other: Replicating Effective Programs
- Replicating Effective Programs (REP) plus coaching (Experimental)
  Interventions: Other: Replicating Effective Programs; Other: Coaching
- Replicating Effective Programs (REP) plus facilitation (Experimental)
  Interventions: Other: Replicating Effective Programs; Other: Facilitation
- Replicating Effective Programs (REP) plus coaching and facilitation (Experimental)
  Interventions: Other: Replicating Effective Programs; Other: Coaching; Other: Facilitation

INTERVENTIONS:
Other: Replicating Effective Programs — Replicating Effective Programs (REP), based on Social Learning Theory and Rogers' Diffusion of Innovations, incorporates program packaging, training, and technical support
Other: Coaching — Coaching is based on the Positive Behavior Interventions and Supports model, addresses staff barriers by building implementers' evidence-based practice (EBP) knowledge, self-efficacy, and skills through clinical support and feedback.
  Arms: Replicating Effective Programs (REP) plus coaching; Replicating Effective Programs (REP) plus coaching and facilitation
Other: Facilitation — Facilitation addresses potential organizational barriers to delivery, including leadership support and acceptance among other staff.
  Arms: Replicating Effective Programs (REP) plus coaching and facilitation; Replicating Effective Programs (REP) plus facilitation

SUMMARY:
In this trial, the investigators will examine the uptake of the evidenced-based IDEAL Goals program, a heart disease risk reduction program, while testing different implementation strategies with our partners in Michigan and Maryland who serve persons with serious mental illness (SMI).

DETAILED DESCRIPTION:
In this trial, the investigators will work with Michigan and Maryland mental health programs to improve the uptake of the 18-month heart disease risk reduction program, IDEAL Goals, to be delivered to persons with SMI enrolled in their behavioral health homes.

ELIGIBILITY:
Community Mental Health Program site staff participants:

Inclusion Criteria

1. Ages 18 and Older
2. English Speaking
3. Agree to complete applicable data collection
4. Agree to engage with the program according to their role (e.g., training, IDEAL Goals program delivery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of IDEAL Goals sessions received by persons with serious mental illness (SMI) at the community mental health program | baseline to 18 months
  Main effects of implementation strategies defined as those who attend sessions that are assigned to the most intensive strategies (Replicating Effective Programs (REP), Coaching, and Facilitation) compared to the least intensive (REP only). The investigators will use electronic health record data on all clients enrolled in the behavioral health home at a participating organization to assess sessions attended. These individuals are not formally enrolled into the trial; their data, obtained under a waiver of informed consent, comprise this outcome.

SECONDARY OUTCOMES:
Number of IDEAL Goals sessions received by persons with serious mental illness (SMI) at the community mental health program | baseline to 18 months
  Marginal effects of implementation strategies defined as those who attend sessions that are assigned to Coaching or Facilitation compared to those not assigned to that same strategy.

OTHER OUTCOMES:
Number of IDEAL Goals sessions received by persons with SMI at the community mental health program at 30 Months (Exploratory) | baseline to 30 months
  Number of sessions received at 30 months
Proportion of visits with recommended tobacco smoking activities (e.g. assessment, counseling if smoker, pharmacotherapy offered if smoker) (Exploratory) | baseline to 18 months, 30 months
Proportion of visits with recommended hypertension activities (e.g. screening, monitoring if have hypertension, medication modification as appropriate) (Exploratory) | baseline to 18 months, 30 months
Proportion of visits with recommended diabetes activities (e.g. screening, monitoring if have diabetes, screening exams if have diabetes, medication modification as appropriate) (Exploratory) | baseline to 18 months, 30 months
Proportion of visits with recommended dyslipidemia activities (e.g. screening, monitoring if have dyslipidemia, medication modification as appropriate ) (Exploratory) | baseline to 18 months, 30 months
Proportion of visits with recommended weight management activities (e.g. counseling) (Exploratory) | baseline to 18 months, 30 months
Self-reported tobacco use among persons with SMI at the community mental health program (Exploratory) | baseline to 18 months, 30 months
  proportion with self-reported tobacco use recorded by staff in electronic health record
Blood pressure (systolic and diastolic) in mmHG among persons with SMI at the community mental health program (Exploratory) | baseline to 18 months, 30 months
HgbA1c level among persons with SMI at the community mental health program. (Exploratory) | baseline to 18 months, 30 months
Lipid values among persons with SMI at the community mental health program (Exploratory) | baseline to 18 months, 30 months
  low density lipoprotein (LDL) mg/dl, high density lipoprotein (HDL) mg/dl,, triglycerides mg/dl, and total cholesterol mg/dl,
BMI (kg/m^2) among persons with SMI at the community mental health program pre and post implementation. (Exploratory) | baseline to 18 months, 30 months
  BMI in kg/m^2 based on measured weight in kg and height in meters
Cardiovascular risk in persons with SMI at community mental health programs (Exploratory) | baseline to 18 months, 30 months
  American Heart Association (AHA) American College of Cardiology Atherosclerotic Cardiovascular Disease (ASCVD) Risk Score, percent risk, higher scores convey more risk
Estimated cost of delivering the IDEAL Goals program and implementation strategies (Exploratory) | baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gail Daumit, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
We will follow NHLBI guidelines.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Yuan CT, Wang NY, Fink T, Almirall D, Appel LJ, Cook C, Cooper LA, Dalcin AT, Gennusa J, Goldsholl S, Kirley E, Liebrecht C, McGinty EE, Smith SN, Terry A, Kilbourne AM, Daumit GL. Achieving cardiovascular health equity in community mental health: study protocol for a cluster-randomized hybrid Type 3 effectiveness-implementation trial. Implement Sci. 2025 Oct 23;20(1):46. doi: 10.1186/s13012-025-01461-4. PMID 41131632